CLINICAL TRIAL: NCT04648254
Title: A Phase 1, Multicenter, Open-label, Dose- Escalation, Safety, Pharmacodynamic, Pharmacokinetic Study of Q702 With a Cohort Expansion at the RP2D in Patients With Advanced Solid Tumors
Brief Title: Oral Axl/Mer/CSF1R Selective Tyrosine Kinase Inhibitor in Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qurient Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q702-ONC-P1-US001
Record Dates: First submitted 2020-11-19; First posted 2020-12-01 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Q702) (Experimental): Participants will receive escalating doses of Q702
  Interventions: Drug: Q702

INTERVENTIONS:
Drug: Q702 — The study drug Q702 will be administered once daily by mouth on Days 1 through 7 and Days 15 through 21 of every treatment cycle.

SUMMARY:
This is a Phase 1, open-label, multicenter, dose-escalation, safety, tolerability, pharmacokinetic and pharmacodynamic study with cohort expansion at the RP2D to evaluate safety and anti- tumor activity of Q702 administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced or metastatic solid tumors, that have progressed following standard of care therapy or for which there is no standard therapy which confers clinical benefit
* Measurable disease per RECIST v 1.1
* ECOG performance status 0 or 1
* Life expectancy of at least 3 months
* Age ≥ 18 years
* Signed, written IRB-approved informed consent form

Exclusion Criteria:

* New York Heart Association Class III or IV cardiac disease, or myocardial infarction, severe unstable angina, coronary/peripheral artery bypass graft, congestive heart failure within the past 6 months
* Have a corrected QT interval (using Fridericia's correction formula) (QTcF) of >470 msec (females) and >450 msec (males)
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Active, poorly controlled autoimmune or inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD), the dose limiting toxicities (DLT) and the safety profile of Q702 | 28 days of cycle 1

SECONDARY OUTCOMES:
Change in the area under curve (AUC) of Q702 | Cycle 1, Days 1,2,8,15,21,22; Cycle 2, Days 1,8,15,22
Change in the maximum plasma concentration (Cmax) of Q702 | Cycle 1, Days 1,2,8,15,21,22; Cycle 2, Days 1,8,15,22
Change in the time of maximum plasma concentration (Tmax) of Q702 | Cycle 1, Days 1,2,8,15,21,22; Cycle 2, Days 1,8,15,22
Tumor response using RECIST version 1.1 throughout study | Baseline up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Atlantic Health System Hospital, Morristown, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jeon Y, Kang H, Yang Y, Park D, Choi B, Kim J, Kim J, Nam K. A Novel Selective Axl/Mer/CSF1R Kinase Inhibitor as a Cancer Immunotherapeutic Agent Targeting Both Immune and Tumor Cells in the Tumor Microenvironment. Cancers (Basel). 2022 Oct 2;14(19):4821. doi: 10.3390/cancers14194821. PMID 36230744